CLINICAL TRIAL: NCT05490680
Title: A Multi-center, Prospective, Randomized, Double-blind, Flexible-dose, Placebo-controlled, Parallel Group Clinical Trial of Sildenafil Oral Film 25 mg, 50 mg, 75 mg and 100 mg for the Treatment of Erectile Dysfunction (ED)
Brief Title: A New Sildenafil Oral Film in Patients With Erectile Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20US-SDF15
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Erectile Dysfunction
Keywords: ED
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo oral film, on-demand use once per day, at maximum 60 films during a 12-week period
  Interventions: Drug: Placebo
- Sildenafil (Experimental): Sildenafil 25 mg, 50 mg, 75 mg or 100 mg oral film (flexible-dose), on-demand use once per day, at maximum 60 films during a 12-week period
  Interventions: Drug: Sildenafil Oral Film 25 mg, 50 mg, 75 mg or 100 mg

INTERVENTIONS:
Drug: Sildenafil Oral Film 25 mg, 50 mg, 75 mg or 100 mg — Sildenafil Oral Film containing 25 mg, 50 mg, 75 mg or 100 mg sildenafil as citrate, flexible-dose
  Other Names: Sildenafil Orodispersible Film
  Arms: Sildenafil
Drug: Placebo — Placebo Oral Film
  Other Names: Placebo-controlled
  Arms: Placebo

SUMMARY:
This is a Phase III, prospective, interventional, multi-center, randomized, double-blind, flexible-dose, placebo-controlled, parallel group clinical study required by FDA to demonstrate the efficacy and safety of Sildenafil oral film 25 mg, 50 mg, 75 mg and 100 mg as compared to placebo in approximately 488 men clinically diagnosed with erectile dysfunction (ED).

DETAILED DESCRIPTION:
The study will consist of a Screening Visit (Visit 0) followed by a 4-week run-in period without treatment and by a Randomization Visit (Visit 1) for the subjects who were compliant in pre-treatment phase. After randomization, the subject will start a 12-week, double-blind, flexible-dose, treatment phase comprising 4 at Site Visits performed 2 weeks after starting the treatment (Visit 2), after additional 2 weeks (Visit 3) and every 4 weeks (Visits 4 and 5) until the End of Study.

The target population for this study is men with ED, including 30-35% of geriatric ED subjects. Subjects < 65 years of age will be randomized to receive the Sildenafil/Placebo oral film at 50 mg dose. Subjects ≥ 65 years of age will be randomized to receive the Sildenafil/Placebo oral film at 25 mg dose. The study foresees a flexible-dose regimen and the starting dosage can be increased to 50 mg (for subjects ≥ 65 years of age), 75 mg or 100 mg dosage, or decreased.

ELIGIBILITY:
Inclusion Criteria:

* Heterosexual male subjects aged ≥18 years;
* Confirmed clinical diagnosis of ED for at least 6 months;
* Involved in a continuous sexual relationship with their partner for at least 3 months.
* Able and willing to provide voluntary written informed consent

Exclusion Criteria:

* Currently suffering from any oromucosal condition or recent oral surgery that could interfere with the study drug;
* Any significant cardiovascular abnormality;
* Patients ≥ 65 years with any degree of hepatic impairment or severe renal impairment or any significant pulmonary, gastrointestinal, hematological, endocrinal, metabolic or neurological disorder;
* Patients < 65 years with severe hepatic impairment;
* Any presence of chronic indwelling urethral catheterization or penile anatomical abnormalities that would significantly impair EF;
* Any history of Peyronie's disease; or who have conditions which may predispose them to priapism;
* Any history or comorbidity of hypoactive sexual desire disorder, premature ejaculation or other ejaculatory disorders or radical prostatectomy;
* Any history of severe/uncontrolled diabetes or radical prostatectomy or spinal cord injury
* Hypersensitivity to Sildenafil or to any of the excipients of the oral film, or idiosyncratic reactions to other PDE5 inhibitors;
* Any history of migraine;
* Any history of complete unresponsiveness to PDE5 inhibitor treatment or significant side-effects with PDE5 inhibitor;
* Subjects with or with history of severe vision impairment, temporary visual disturbances (blurred vision, increased light sensitivity and color change), retinitis pigmentosa, Non-Arteritic Anterior Ischemic Optic Neuropathy (NAION) or any optic neuropathy;
* Subjects taking a strong CYP3A4 inhibitor(s);
* During the course of the study, subjects are not allowed to take any prescription, over-the-counter, herbal, or naturopathic products for "male enhancement" or the treatment of ED;
* During the course of the study, subjects are not allowed to take any form of nitric oxide donors such as organic nitrates or organic nitrites either regularly and/or intermittently, and guanylate cyclase (GC) stimulators;
* Patients must be stable on therapy with Alpha-blockers or Amlodipine at inclusion and already taking a PDE5 inhibitor without any safety concern prior to initiating the study (i.e., no history of significant side-effects with co-administration of PDE5 inhibitors);
* Subjects known to abuse alcohol or drugs that could interfere with the patient's safety or study compliance
* Subjects who are illiterate or are unable to understand how to use eDiary and complete the questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Safety of Sildenafil doses versus placebo | 12 weeks of treatment
  Safety of Sildenafil doses versus placebo, i.e., the proportion of subjects with at least one Treatment Emergent Adverse Events (TEAEs) of Special Interest ("Headache" or "Dizziness")
Efficacy of Sildenafil doses versus placebo - IIEF-EF | Baseline to the end of the 12-week treatment period
  Efficacy of Sildenafil oral film versus placebo evaluated using co-primary efficacy endpoint from the change in Erectile Function (EF) domain of the International Index for Erectile Function (IIEF) questionnaire
Efficacy of Sildenafil doses versus placebo - SEP Question 2 | Between the 4-week pre-treatment period and the end of the 12-week treatment period
  Efficacy of Sildenafil oral film versus placebo evaluated using co-primary efficacy endpoint from the change in percentage of "yes" responses to Sexual Encounter Profile (SEP) Question 2
Efficacy of Sildenafil doses versus placebo - SEP Question 3 | Between the 4-week pre-treatment period and the end of the 12-week treatment period
  Efficacy of Sildenafil oral film versus placebo evaluated using co-primary efficacy endpoint from the change in percentage of "yes" responses to SEP Question 3

SECONDARY OUTCOMES:
Safety TEAE of special interest - headache | Over 12 weeks of treatment as compared to placebo
  The incidence of TEAEs of Special Interest of headache
Safety TEAE of special interest - dizziness | Over 12 weeks of treatment as compared to placebo
  The incidence of TEAEs of Special Interest of dizziness
Safety TEAE of vasomotor drug effects | Over 12 weeks of treatment as compared to placebo;
  The incidence of TEAEs that may be suggestive of vasomotor drug effects and the proportion of subjects with at least one of these TEAEs

OTHER OUTCOMES:
Exploratory efficacy of Sildenafil oral film compared to placebo - attempts | Up to 12 weeks of treatment
  Number of attempts for sexual intercourse
Exploratory efficacy of Sildenafil oral film compared to placebo - overall treatment satisfaction | Up to 12 weeks of treatment
  Mean treatment satisfaction as assessed by Overall Treatment Satisfaction score on a 5-point scale (4=excellent; 3=good; 2=fair; 1=poor; 0=none)
Exploratory efficacy of Sildenafil oral film compared to placebo - GAQ | Up to 12 weeks of treatment
  Proportion of subject responses to Global Assessment Questionnaire (GAQ) consisting of 2 questions (Yes or No): Question 1 'Has the treatment you have been taking improved your erectile function?' and if necessary, Question 2 'If yes, has the treatment improved your ability to engage in sexual activity?'.
Exploratory efficacy of Sildenafil oral film compared to placebo - drug product palatability | Up to 12 weeks of treatment
  Subjective measures of the Drug Product Palatability consisting of 5 specific questions: "1. Rate the oral sensation/mouthfeel of the drug product"; "2. Rate the taste of the drug product"; "3. How strong is the taste?"; "4. Rate the aftertaste of the drug product"; and "5. How strong is the aftertaste?". For questions 1, 2, and 4, the range of responses is: "very unpleasant, unpleasant, no sensation/mouthfeel, pleasant, very pleasant." For questions 3 and 5, the range of responses is: "very strong, strong, moderate, mild, no taste".

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D. Efros, MD, Principal Investigator — Accumed Research Associates
Locations (18):
- United States (18):
  - G & L Research LLC., Foley, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Arkansas Urology Research Center, Little Rock, Arkansas
  - Urology Group of Southern California, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Innovation Medical Group LLC (Endo Care of South Florida), Fort Lauderdale, Florida
  - Clintex Research Group, Miami, Florida
  - Coral Research Clinic, Miami, Florida
  - Harmony Clinical Research, North Miami Beach, Florida
  - Innovation Clinical Trials: Medical Reseach Center, Palmetto Bay, Florida
  - Precision Clinical Research, LLC, Sunrise, Florida
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - AccuMed Research Associates, Garden City, New York
  - Rochester Clinical Research, Inc, Rochester, New York
  - Alliance for Multispeciaty Research, LLC, Knoxville, Tennessee
  - Mt. Olympus Medical Research Group, LLC, Sugar Land, Texas
  - Tranquil Clinical and Research Consulting Services, LLC, Webster, Texas
  - Virginia Urology, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No